CLINICAL TRIAL: NCT02018809
Title: Using Social Support To Improve Medication Adherence In Statin Users With Diabetes
Brief Title: Social Forces to Improve Statin Adherence (Study A)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 819129-A
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Medication Adherence; High Blood Pressure; Diabetes
Keywords: Medication Adherence; High Blood Pressure; Diabetes; Statins
MeSH Terms: conditions — Medication Adherence; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MAP Daily Notification (Experimental): The subject's MAP receives daily notification about whether subject took statin.
  Interventions: Behavioral: Medication Adherence Partner; Device: Electronic pill bottle
- MAP Weekly Notification (Experimental): The subject's MAP receives weekly about how often the subject took statin during previous week.
  Interventions: Behavioral: Medication Adherence Partner; Device: Electronic pill bottle
- MAP Missed Doses (Experimental): The subject's MAP receives notification if the subject missed >2 consecutive daily doses of statin.
  Interventions: Behavioral: Medication Adherence Partner; Device: Electronic pill bottle
- Usual Care (Other): Usual care with GlowCap.
  Interventions: Device: Electronic pill bottle

INTERVENTIONS:
Behavioral: Medication Adherence Partner
  Arms: MAP Daily Notification; MAP Missed Doses; MAP Weekly Notification
Device: Electronic pill bottle — This device can remotely track medication taking and will be used by subjects to store once-a-day statin medication already prescribed pre-trial.
  Other Names: Vitality GlowCap

SUMMARY:
To assess the effectiveness of reporting statin adherence patterns to a Medication Adherence Partner (MAP) in improving the outcome of statin adherence versus usual care as measured by an electronic pill bottle.

Hypothesis: Subjects with a MAP receiving daily adherence feedback will have the highest statin adherence of any arm, as measured by pill bottle data.

DETAILED DESCRIPTION:
We propose to complete a randomized controlled trial (RCT) of 200 subjects with medication treated diabetes and evidence of poor adherence to a statin medication (<70% medication possession ratio determined through pharmacy records; no combination meds). Study subjects will use an electronic pill bottle (GlowCap) to store their statin medication. Study subjects will identify potential Medication Adherence Partners (MAPs) who can receive information about their adherence patterns at enrollment. For the 90-day trial, subjects will be randomized to: 1) the subject's MAP receives daily notification about whether subject took statin; 2) the subject's MAP receives weekly about how often the subject took statin during previous week; 3) the subject's MAP receives notification if the subject missed >2 consecutive daily doses of statin; and 4) usual care (GlowCaps without any notifications). The primary outcome will be the percent of statin doses taken during the study as measured by the GlowCaps. The secondary outcome will be subjects' statin medication possession ratio (MPR) during the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is Humana insured
* The subject is an English speaking adult
* Age range ≥18 years
* The subject has diagnosis with diabetes for ≥12 months
* The subject has an MPR <70% to a statin medication
* Subject denies side-effects to their statin medication
* The subject identified a person who agreed to serve as their MAP

Exclusion Criteria:

* The subject is <18 years old
* The subject is considered part of a vulnerable population (is a prisoner, a cognitively impaired person, or a pregnant woman)
* On statin combination medication
* The subject does not identify an individual who agrees to serve as their MAP
* The subject reports a clinically important side effect to the statin medication or active liver disease:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Reese, MD, MSCE, Principal Investigator — UPenn PSOM; Judd B Kessler, PhD, Principal Investigator — UPenn, Wharton; Kevin Volpp, MD, PhD, Principal Investigator — UPenn, PSOM
Locations (1):
- University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MAP Daily Notification: The subject's MAP receives daily notification about whether subject took statin.
  Medication Adherence Partner
  Electronic pill bottle: This device can remotely track medication taking and will be used by subjects to store once-a-day statin medication already prescribed pre-trial.
- MAP Weekly Notification: The subject's MAP receives weekly about how often the subject took statin during previous week.
  Medication Adherence Partner
  Electronic pill bottle: This device can remotely track medication taking and will be used by subjects to store once-a-day statin medication already prescribed pre-trial.
- MAP Missed Doses: The subject's MAP receives notification if the subject missed >2 consecutive daily doses of statin.
  Medication Adherence Partner
  Electronic pill bottle: This device can remotely track medication taking and will be used by subjects to store once-a-day statin medication already prescribed pre-trial.
Period: Overall Study
Arm/Group | MAP Daily Notification | MAP Weekly Notification | MAP Missed Doses | Usual Care
Started | 50 | 50 | 50 | 50
Completed | 50 | 50 | 50 | 50
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MAP Daily Notification | MAP Weekly Notification | MAP Missed Doses | Usual Care | Total
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10) | 66 (10) | 65 (9) | 67 (10) | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 22 | 23 | 100
  Male | 20 | 25 | 28 | 27 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 2 | 1 | 12
  Not Hispanic or Latino | 46 | 45 | 48 | 49 | 188
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 3 | 4 | 3 | 10
  White | 45 | 41 | 43 | 45 | 174
  More than one race | 5 | 4 | 0 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Statin Adherence
Description: The primary outcome will be the percent of statin doses taken during the study as measured by the GlowCaps.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: percentage of correct statin doses
Arm/Group | MAP Daily Notification | MAP Weekly Notification | MAP Missed Doses | Usual Care
Number analyzed (Participants) | 50 | 50 | 50 | 50
percentage of correct statin doses | 86 (.18) | 85 (.20) | 86 (.17) | 85 (.15)

2. Secondary Outcome: Morisky Medication Adherence Scale (MMAS)
Description: The secondary outcome will be subjects' self-reports medication adherence. Morisky et al. developed this 8-item MMAS (MMAS-8) in 2008. The first seven items are Yes/No responses while the last item is a 5-point Likert response. The scoring scheme is: "Yes" = 0 and "No" = 1 (and "0" = 0 and "1-4" = 1 for Likert question). The items are summed to give a range of scores from 0 to 8. Respondents' summed score get grouped as follows: "0" = High Adherence; "1-2" = Medium Adherence; "3-8" = Low Adherence.
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | MAP Daily Notification | MAP Weekly Notification | MAP Missed Doses | Usual Care
Number analyzed (Participants) | 50 | 50 | 50 | 50
units on a scale | 5.38 [4 to 6.75] | 6 [4.75 to 7] | 5.75 [4.75 to 7] | 5.75 [4.75 to 7]

ADVERSE EVENTS:
Arm/Group | MAP Daily Notification | MAP Weekly Notification | MAP Missed Doses | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
The interventions lasted only 3 months; differences in adherence might emerge over a longer period of time. The primary outcome of pill-bottle-measured adherence has limitations, including bottle malfunction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No